CLINICAL TRIAL: NCT04218019
Title: Effect of Timing of Tumor-Treating Fields Plus Short-Course Radiation in Elderly Patients With Glioblastoma
Brief Title: Effect of Timing of Tumor-Treating Fields Plus Short-Course Radiation
Acronym: GERAS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Organizational reasons
Sponsor: Juergen Debus (Other)
Responsible Party: Sponsor-Investigator, Juergen Debus, Head of Department, University Hospital Heidelberg
Organization: University Hospital Heidelberg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GERAS
Record Dates: First submitted 2020-01-02; First posted 2020-01-06 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Newly Diagnosed Glioblastoma in Patients ≥70 Years

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Tumor Treating Fields (TTFields, Optune®) treatment (Experimental): TTF will be started together with hypofractionated radiotherapy (+/- 5 days) with or without Temozolomide (according to the standard and local physician's decision). Chemoradiotherapy with temozolomide and hypofractionated radiotherapy is regarded as standard therapy and not part of the intervention. In case of chemoradiotherapy temozolomide will be applied according to the standard of the participating trial center. Use of antiemetic and infection prophylaxis will be at the discretion of the investigator.
  Interventions: Device: TTFields
- Late TTF treatment (Active Comparator): Patients will be treated with hypofractionated radiotherapy with or without temozolomide (according to the local standard and physician's decision). Radiotherapy and treatment with temozolomide is regarded as standard therapy and not part of the intervention. In case of chemoradiotherapy temozolomide will be applied according to the standard of the participating trial center. Use of antiemetic and infection prophylaxis will be at the discretion of the investigator. Late TTFields treatment will start 4 weeks after the end of radiotherapy.
  Interventions: Device: TTFields

INTERVENTIONS:
Device: TTFields — The NovoTTF-200 A device used in this trial delivers very low intensity, alternating electric fields to the tumor site through the scalp. These fields are known as Tumor Treating Fields or TTFields.

SUMMARY:
The purpose of the study is to assess timing of TTFields use as well as safety, feasibility and preliminary efficacy of treatment with TTFields in elderly patients with newly diagnosed GBM simultaneous to RT/ CRT.

The primary aim of the trial is to establish a safely conducted therapy rate higher than 0.8 in the treatment arm.

DETAILED DESCRIPTION:
Despite the immense effort made over the years with different treatment modalities, the survival of patients with newly diagnosed GBM is still very poor; no treatment is curative; and the quality of life of patients with this tumor is compromised significantly, not only by their disease but also by side effects of these rigorous treatment plans. Especially in elderly patients, a treatment modality is needed that will improve the results of current standard treatments without further impairing the quality of life of these patients for their limited life span.

The objective is to test the feasibility and timing of treatment with the TTFields device in elderly patients with newly diagnosed GBM simultaneous or subsequent to RT/ CRT.

The primary rationale to conduct this study is to improve treatment in the segment of high-grade brain tumors with the highest medical need.

All procedures regarding TTFields are representing routine clinical care within the approved use of the medical product in Germany; the present trial aims to investigate the optimal timing of TTFields use in elderly GBM patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, newly diagnosed glioblastoma (astrocytoma WHO grade IV)
* Indication for hypofractionated radiotherapy or hypofractionated chemo-radiotherapy with temozolomide
* Open biopsy or resection
* Craniotomy or intracranial biopsy site must be adequately healed
* Informed consent
* Age: >65 years
* KPS ≥50%
* Ability of subject to understand character and individual consequences of the clinical trial
* Written informed consent of participation

Exclusion Criteria:

* Concurrent participation in another competing interventional clinical trial studying a drug or treatment regimen.
* Any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol requirements and/or follow-up procedures; those conditions should be discussed with the patient before trial entry
* Prior RT of the brain
* Patients who have not yet recovered from acute high-grade toxicities of prior therapies
* MRI or TTFields contraindication (e.g. cardiac pacemaker, implanted defibrillator, certain cardiac valve replacements, certain metal implants, patients with severe skull defects such as a missing bone flap, programmable shunts)
* Known hypersensitivity to conductive hydrogels
* Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Safely conducted therapy rate (SCTR) | at least one week of treatment
  The proportion of patients fulfilling the inclusion/exclusion criteria who were treated for at least one week according to protocol and neither experienced neither NCI-CTC-AEs of Grade 3 nor 4
Number of participants with treatment related adverse events as assessed by CTCAE V 5.0. | within 31 weeks after treatment
  Safety and tolerability of TTFields Treatment combined with radiotherapy/chemo-radiotherapy

SECONDARY OUTCOMES:
Progression-free survival | within 6 month after treatment
  according to RANO criteria
The correlation between the Optune device usage and the health-related quality of life of elderly patients and families undergoing this therapy in combination with radiotherapy/chemo-radiotherapy. | within 31 weeks after treatment
  Score on the EORTC QoL C15-Pal
The correlation between the Optune device usage and the health-related quality of life of elderly patients and families undergoing this therapy in combination with radiotherapy/chemo-radiotherapy. | within 31 weeks after treatment
  Score on the EORTC QoL BN20

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Debus, Prof., Principal Investigator — Head of Department
Locations (1):
- University Hospital of Heidelberg, Radiation Oncology, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No